CLINICAL TRIAL: NCT03197480
Title: Identifying Ocular and Systemic Biomarkers for Response to Aflibercept in Asian Patients With Centre Involving Diabetic Macular Edema: A Prospective Clinical Trial
Brief Title: Diabetic Macular Edema Asian Response (DEAR) Study: Biomarkers for Response to Aflibercept in Asian Patients With Center Involving DME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Santen Pharmaceutical Co., Ltd. (Industry); Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1436/19/2017
Record Dates: First submitted 2017-06-05; First posted 2017-06-23 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Macular Edema
Keywords: Anti-Vascular Endothelial Growth Factor; Aflibercept; Intravitreal injection; Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: This is a prospective observational clinical trial with only the use of a standard care of drug, aflibercept. All study eyes will receive intravitreal aflibercept at the initial injection and x 4 monthly injections including at month 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DME treatment group (Other): All patients will received 4 intravitreal injections of aflibercept.
  Based on the OCT outcome they will be classified into 2 groups for assessment of biomarkers:
  Less than 20% reduction in CRT on OCT or <5 letter improvement of VA (if VA<6/6 and CRT>=340) Rapid (Mac Dry at M4) Delayed: Persistent fluid at M4, but more than 20% reduction in CRT on OCT
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — All subjects will receive 4 monthly intravitreal injections of aflibercept

SUMMARY:
To investigate whether ocular imaging and proteomic biomarkers; and systemic biochemical, metabolomic, and genetic biomarkers predict treatment response to intravitreal aflibercept in a cohort of patients with DME.

DETAILED DESCRIPTION:
This is a prospective observational clinical trial with only the use of a standard care of drug, aflibercept. All study eyes will receive intravitreal aflibercept at the initial injection and x 4 monthly injections including at month 3.

ELIGIBILITY:
Inclusion Criteria:

Participant

1. Age >=21 years
2. Diagnosis of Diabetes Mellitus (Type 1 or type 2)

   1. Current regular use of insulin or oral hypoglycemic agents for treatment of diabetes
   2. Documented diabetes by ADA and/or WHO criteria.
3. Able and willing to provide informed consent.

Study Eye

1. Best corrected ETDRS visual acuity score <= 78 (ie 20/32 or worse)
2. On Clinical Examination, definite retinal thickening due to diabetic macular edema involving the center of the macula.
3. Diabetic macular edema present on OCT (central subfield thickness on OCT >=300um with spectralis (Heidelberg)
4. Media clarity, pupillary dilation and individual cooperation sufficient for study procedure including fundus photography.

Exclusion Criteria:

Participant

1. End stage renal failure requiring hemodialysis or peritoneal dialysis.
2. Medical condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
3. Participation in an investigational trial within 30 days of enrolment which involves treatment with unapproved investigational drug
4. Known allergy to any component of the study drug.
5. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110 on repeated measurements). If blood pressure is brought below 180/110 by anti-hypertensive treatment, individual can become eligible.
6. Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization.
7. Systemic anti-VEGF or pro-VEGF treatment within three months prior to randomization or anticipated use during the study.
8. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 24 months. Women who are potential study participants should be questioned about the potential for pregnancy.
9. Patient with non study eye VA: counting finger or worse (i.e. only one seeing eye) will be excluded.

Study Eye

1. Macular edema is considered to be due to a cause other than diabetic macular edema. An eye should not be considered eligible if: (1) the macular edema is considered to be related to ocular surgery such as cataract extraction or (2) clinical exam and/or OCT suggest that vitreoretinal interface abnormalities (e.g., a taut posterior hyaloid or epiretinal membrane) are the primary cause of the macular edema.
2. An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition).
3. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.)
4. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by more than three lines (i.e., cataract would be reducing acuity to worse than 20/40 if eye was otherwise normal).
5. History of an anti-VEGF treatment for DME in the past 3 months or history of any other treatment for DME at any time in the past 3 months (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids).
6. History of pan-retinal photocoagulation within 3 months prior to randomization or anticipated need for immediate pan-retinal photocoagulation. (eg. Proliferative diabetic retinopathy. Cases with severe non-proliferative diabetic retinopathy will still be eligible)
7. History of ocular anti-VEGF treatment for a disease other than DME in the past 3 months
8. History of major ocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior four months or anticipated within the next six months following randomization.
9. History of YAG capsulotomy performed within two months prior to randomization.
10. Aphakia.
11. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.
12. History of intravitreal steroids within the last 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
CRT | 12 Months
  Mean change in Central Retinal Thickness

SECONDARY OUTCOMES:
BCVA | 12 Months
  Mean change in Best Corrected Visual Acuity
Change in vascular density by OCTA | Baseline, Month 12
  Change in vascular density by OCTA in different layer
Percentage of patients with a BCVA improvement of 15 letters or more | Baseline, Month 12
  Percentage of patients with a BCVA improvement of 15 letters or more
Percentage of patients with a BCVA improvement of 10 letters or more | Baseline, Month 12
  Percentage of patients with a BCVA improvement of 10 letters or more
Mean BCVA at each injection number | 12 Months
  Mean BCVA at each injection number
Mean change in BCVA across all the study injection numbers | Baseline, Month 12
  Mean change in BCVA across all the study injection numbers
Percentage of patients with BCVA improvement | Baseline, Month 12
  Percentage of patients with BCVA improvement
Percentage of BCVA losers | Baseline, Month 12
  Percentage of BCVA losers
Percentage of patients improving to 20/40 or better | Baseline, Month 12
  Percentage of patients improving to 20/40 or better

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Tan, Study Director — Singapore National Eye Center
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03197480/Prot_SAP_000.pdf